CLINICAL TRIAL: NCT04730648
Title: Acute Myocardial Infarction and Unstable Angina Patients With PCSK9 Inhibitor Usage Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Ying Li, professor, Shenzhen People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Among-Us study
Record Dates: First submitted 2020-11-26; First posted 2021-01-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Lipid Metabolism; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pcsk9 inhibitor group (Experimental): patients with severe coronary stenosis diagnosed ACS. The baseline blood and urine would be collected, thereafter, the PCSK9 inhibitor would be injected. 64-72 hours after, the blood and urine sample collection would be performed.
  Interventions: Drug: PCSK9 inhibitor
- control group (No Intervention): Patients with comparable age, sex ratio, and BMI, but coronary arteries are relatively normal evaluated by coronary angiography. their blood and urine would be collected as the control group.

INTERVENTIONS:
Drug: PCSK9 inhibitor — For newly diagnosed ACS patients with diabetes, multivessel occlusion, or recurrent ACS attack, who are willing to accept PCSK9 inhibitor injection.
  Arms: pcsk9 inhibitor group

SUMMARY:
Acute coronary syndrome (ACS) is a lethal disease, reduced low-density lipoprotein (LDL) cholesterol due to inhibition of proprotein convertase subtilisin/kexin 9 (PCSK9) reduces cardiovascular events and improve cardiovascular prognosis. we assuming that PCSK9 inhibitor could bring metabolic change in serum, in order to investigate the metabolic modification, we conduct this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis ACS patient by serum biomarker and coronary arteriography.

Exclusion Criteria:

* Severe renal dysfunction acute or chronic bacterial and viral infections sleep apnea cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2023-04-23 (Estimated)

PRIMARY OUTCOMES:
cardiovascular prognosis | 52 weeks
  composite outcome of time to first occurrence of cardiovascular death, myocardial infarction, unstable angina and heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Tangzhiming Li, PhD., Principal Investigator — Department of Cardiology, Shenzhen People's Hospital, Shenzhen 518020, Guangdong, China
Locations (1):
- Tangzhiming Li, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Ou Z, Yu Z, Liang B, Zhao L, Li J, Pang X, Liu Q, Xu C, Dong S, Sun X, Li T. Evolocumab enables rapid LDL-C reduction and inflammatory modulation during in-hospital stage of acute coronary syndrome: A pilot study on Chinese patients. Front Cardiovasc Med. 2022 Aug 9;9:939791. doi: 10.3389/fcvm.2022.939791. eCollection 2022. PMID 36017088